CLINICAL TRIAL: NCT03603236
Title: Evaluation of the Possible Relationship Between Preeclampsia and Periodontal Disease With Clinical Periodontal, Biochemical and Microbiological Data
Brief Title: Evaluation of the Possible Relationship Between Preeclampsia and Periodontal Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Recep Tayyip Erdogan University Training and Research Hospital (Other)
Collaborators: Ege University (Other)
Responsible Party: Principal Investigator, Gul Yildiz Telatar, Principal Investigator, Recep Tayyip Erdogan University Training and Research Hospital
Other Study IDs: 40465587-28
Record Dates: First submitted 2018-07-17; First posted 2018-07-27 (Actual); Last update posted 2018-07-27 (Actual); Status verified 2018-07

CONDITIONS: Preeclampsia; Periodontal Disease
MeSH Terms: conditions — Pre-Eclampsia; Periodontal Diseases | interventions — Blood Specimen Collection; Urinalysis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Tissue samples from four centers will be taken from the maternal and fetal surfaces of the placenta Saliva samples of pregnant women
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- preeclampsia: 18-40 aged diagnosed with preeclampsia
  Interventions: Diagnostic Test: preeclampsia; Diagnostic Test: control
- control: 18- 40 aged healthy females over 37. weeks of pregnant with no history of preeclampsia
  Interventions: Diagnostic Test: preeclampsia; Diagnostic Test: control

INTERVENTIONS:
Diagnostic Test: preeclampsia — liver function tests, kidney function tests and platelets measures the ratio of protein to creatinine
  Other Names: blood sample, urine test
Diagnostic Test: control — liver function tests, kidney function tests and platelets measures the ratio of protein to creatinine
  Other Names: blood sample, urine test

SUMMARY:
The primary objective of the study is to assess the incidence and severity of the periodontal infection of patients with preeclampsia.

The secondary objective of the study is to analyze the relationship between preeclampsia and periodontal infection, using clinical, biochemical and microbiological methods.

DETAILED DESCRIPTION:
Preeclampsia is identified as an important cause for mother and newborn mortality. Inspite of extensive research, the exact etiological relations have not been established.

Periodontal disease is a subclinical and persistent infection source which induces the systemic inflammatory reactions and increases the risk of preeclampsia. It is believed that the results will set light to the etiology of preeclampsia and will help to develop strategies to prevent the disease.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women with preeclampsia
* 37. weeks of pregnant women with no history of preterm labor

Exclusion Criteria:

* Genitourinary infection,
* pregnancy or pre-pregnancy hypertension,
* HIV infection,
* diabetes mellitus,
* multiple pregnancy, preterm labor / low birth weight,
* smoker and alcohol use history,
* IVF pregnancy,
* placental, cervical and uterine anomalies,
* pregnancy with intrauterine growth retardation,
* pregnancies with congenital or chromosomal fetal anomalies,
* significant vaginal bleeding,
* infertility stories,
* drug addicts,
* poor socioeconomic level

Ages: 21 Years to 34 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — pregnant women
Study Population: The study is planned to be a case-control study. Workgroup consists of 50 patients which diagnosed with preeclampsia between the age of 18 and 40. Control group consists of healthy females over 37. weeks of pregnant with no history of preeclampsia.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-02-17 (Actual); Primary Completion 2018-09-17 (Estimated); Study Completion 2018-12-15 (Estimated)

PRIMARY OUTCOMES:
prostaglandin E2 | 1 Day
  prostaglandin E2 levels will be evaulated in salivary, serum and placenta samples using ELISA test Normal value:29-97 pg / ml
TNF-Alpha (Tumor necrosis factor -Alpha) | 1 day
  TNF-Alpha levels will be evaulated in salivary, serum and placenta samples using ELISA test Normal value:42-203pg/ml
IL-1beta (Interleukin 1 beta) | 1 day
  IL-1beta levels will be evaulated in salivary, serum and placenta samples using ELISA test Normal value:3-227pg/ml

SECONDARY OUTCOMES:
Porphyromonas gingivalis | 1 Day
  Presence of Porphyromonas gingivalis will be checked by rPCR method. Score 1: Present Score 2: None Tannerella Forsythia (+,-)
Tannerella Forsythia | 1 Day
  Presence of Tannerella Forsythia will be checked by rPCR method. Score:1 Present. Score 2: None

CONTACTS AND LOCATIONS:
Overall Officials: Gül Yıldız Telatar, Principal Investigator — Recep Tayyip Erdogan University Dentistry Faculty; Önder Gürlek, Dr., Principal Investigator — Ege University
Locations (5):
- Turkey (Türkiye) (4):
  - Ege University Dentistry Faculty, Izmir
  - İzmir Health Sciences University, Tepecik Training and Research Hospital Department of Obstetrics and Gynecology, Izmir
  - Recep Tayyip Erdogan University Dentistry Faculty, Rize
  - Recep Tayyip Erdogan University Faculty of Medicine, Rize
- Glaskow Dental School , School of Medicine University of Glasgow, Glaskow, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Data will be available within 6 months of study completion

REFERENCES:
- [Background] Jaiman G, Nayak PA, Sharma S, Nagpal K. Maternal periodontal disease and preeclampsia in Jaipur population. J Indian Soc Periodontol. 2018 Jan-Feb;22(1):50-54. doi: 10.4103/jisp.jisp_363_15. PMID 29568173
- See also: Maternal periodontal disease and preeclampsia in Jaipur population. — http://www.ncbi.nlm.nih.gov/pubmed/29568173